#### NCT# 014466972

## UNIVERSITY OF CALIFORNIA, SAN FRANCISCO CONSENT TO PARTICIPATE IN A RESEARCH STUDY

Study Title: CC#117513: Reversing Hormone Resistance in Advanced Breast Cancer with Pazopanib

This is a clinical trial, a type of research study. Your study doctor, Hope Rugo, MD and/or her associates from the UCSF Helen Diller Family Comprehensive Cancer Center will explain the clinical trial to you.

Clinical trials include only people who choose to take part. Please take your time to make your decision about participating. You may discuss your decision with your family and friends and with your health care team. If you have any questions, you may ask your study doctor.

You are being asked to take part in this study because you have metastatic breast cancer (breast cancer that has spread to other parts of the body) that is known to be estrogen and/or progesterone receptor positive and your cancer has progressed while on hormone treatment.

## Why is this study being done?

The purpose of this study is to find out what effects, good and/or bad, of adding pazopanib (the study drug) to your current hormonal treatment (you may take either anastrozole [Arimidex] or letrozole [Femara]). The study will see whether the combination is safe and easy to tolerate. If your study doctor is able to detect tumor cells in your blood before the treatment and/or during the treatment, he/she will also monitor the change of these tumor cells.

Pazopanib is a drug taken by mouth that belongs to a class of medications called tyrosine kinase inhibitors. It works by slowing or stopping new blood vessel growth that can feed cancer growth. It has been approved by the United States Food and Drug Administration (FDA) for the treatment of advanced kidney cancer and certain types of advanced soft tissue sarcoma, but is not approved in the treatment of breast cancer. Thus, its use in this study is considered investigational.

This study is being coordinated by UCSF. The makers of pazopanib, Novartis Pharmaceuticals, are providing funding necessary for trial conduct and some study related tests.

## How many people will take part in this study?

This study will be conducted at UCSF. Up to 30 patients will be enrolled in this study.

## What will happen if I take part in this research study?

This study will enroll participants in two-steps. Initially, 14 patients will be enrolled. If at least 1 patient shows that he/she is benefiting clinically from the study drug, then the study will proceed

PAGE 1 OF 19

to the second step. At the second step, 13-16 more patients will be enrolled. The study doctor will let you know which step of the study you will be enrolling in.

If you decide to participate in this study, you will need to have several tests done to make sure that you qualify for this study. If you are eligible to participate in the study, you will enter the treatment phase of the study.

## Before you begin the main part of the study...

You will need to have the following exams, tests or procedures to find out if you can be in the study. Some of these exams, tests or procedures are part of regular cancer care and may be done even if you don't join the study. Some exams, tests, and procedures are being done because they are a part of the study. These are indicated as "study tests". If you had some of them recently (within 3 weeks before the study begins), they may not need to be repeated. This will be up to your study doctor. The screening visit to complete all of the tests and procedures listed below will take approximately 2-3 hours.

- Physical examination (including your height and weight)
- Medical history (including a review of your prior and current medications)
- Vital signs (heart rate, blood pressure, temperature)
- Electrocardiogram (ECG) An ECG records the natural electrical activity of your heart. You will lie down, and wires or "leads" will be attached to your chest with an adhesive. You will be asked to lie still while the machine prints out an electrical "picture" of your heart activity. The ECG takes about 15 minutes.
- Blood tests: a small sample of blood (about 11 teaspoons) for the following:
  - o Routine blood tests to measure your blood counts, and kidney, liver, and thyroid function.
  - For research purposes to check for circulating tumor cells (very small numbers of cancer cells in the blood) study test
  - o To check your immune system study test
- A urine sample will be collected to check for protein study test
- Tumor assessments (CT or MRI of the chest, abdomen and pelvis if you have disease that can be measured, or a Bone Scan or PET/CT if you have cancer in the bones)
  - CT scan: A CT scan uses special x-ray equipment to make detailed pictures of body tissues and organs. For the CT scan, you may be given a "contrast material" (a special dye that makes it easier for doctors to see different tissues in your body). The contrast material may be given orally, intravenously, or rectally (less likely). Oral contrast material is given to you to drink and is used to help outline the stomach and intestines. Intravenous (IV) contrast material is given to you by injecting the contrast material into a line which is attached to a needle in your arm, and is used to get clearer pictures of your body cavity. A rectal contrast fills up the loops of your lower bowel so the doctors can see your tumor better. After you have been given the contrast material (either by mouth, by vein, or rectum), you will lie flat on a table that will move you into the CT scan machine. You will be asked to lie still and may be asked to hold your breath for

a few seconds. The CT scan is done in the radiology department and takes about half an hour.

- MRI scan: An MRI scan takes an image of your body to observe the location and size of your tumor. When having an MRI (Magnetic Resonance Imaging) scan, you will lie still on a table that slides into a tunnel slightly wider than your body. People who feel uncomfortable in confined spaces (claustrophobia) may feel uncomfortable in the narrow cylinder. MRIs use powerful magnets to make images. Therefore, persons with certain metal implants, such as pacemakers should not have an MRI (If you have an implant or any metal in your body, please check with your study care doctor to know whether you can have an MRI or not.) For people without metal implants, there are no known health risks associated with exposure to the magnet. As images are taken, a loud banging noise will be produced. Earplugs will be available if needed. The MRI can be stopped at any time at your request. You will lie there quietly for about one hour, during which time you will hear a loud machine-like noise. The MRI scan is done in the radiology department and takes approximately an hour and a half to complete.
- PET/CT scan: A PET/CT scan is a special type of test to show how the organs and cells work in your body and is done to show activity of the cells in your tumor. Your scan will begin with an injection of a radioactive substance into a vein in your arm. You will be asked to rest quietly for a period of time (usually about 20 to 40 minutes) as the radioactive substance circulates throughout your body. After this time, you will be positioned within a large ring (similar to a big donut hole) on a scanning bed. Once positioned properly, the bed will move you into the scanner. As pictures are being taken, you will be asked to remain very still so clear images will be taken. The imaging time takes about one hour.
- Bone scan: a bone scan is a test to find areas of increased or decreased bone cell metabolism. Metabolism is the process of tissue cells dying and being replaced by new cells. A bone scan may be performed before you start the treatment if you have cancer cells in the bone if you have not had a PET scan.
- Leftover tumor tissue collection study test

The researchers will obtain a sample of leftover tumor tissue from any biopsy or surgery you may have as part of your regular cancer care if available. This tissue will be used to look for changes (mutations) in genes (DNA) and tumor markers (substances produced by your body in response to cancer).

• Tumor Biopsy – *Optional* – study test. A doctor will remove a piece of your tumor tissue if it can be obtained. This is called a biopsy. Usually, this biopsy involves the use of a small needle which is directed into your tumor site with the guidance of an imaging machine such as a CT scan or a Doppler ultrasound, if necessary. Your tumor sample will be used to help us understand the possible mutations your cancer cells may have. This



procedure takes about 30 minutes. You will sign a separate consent page for this procedure. Your treating physician will determine if this procedure is safe for you to have.

## During the main part of the study...

If the exams, tests and procedures show that you can be in the main part of the study, and you choose to take part, then you will need the following tests and procedures. They are part of regular cancer care.

If you agree to take part in this study, it is very important that you tell your study doctor before starting on this study about all of the medicines you are taking (over-the-counter medications, supplements, prescription medications, or illegal drugs) including any medicines you have taken within the past 2 weeks. This is important because some medicines can change the way your body handles other medicines and this can increase the risk of side effects. In addition, please talk with the study doctor before you begin taking any new medications or supplements during this study.

Your study doctor will look at the medicines you are currently taking to make sure you are allowed to take them on the study. You may be asked to change some of the medicines you are taking. If you need to take a medicine that is not allowed and it cannot be replaced with another medicine, you will not be asked to stop taking it; however, you will not be able to take part in this study.

While you are participating in this study, you will come to the clinic every 2 weeks for the first 4 weeks. After that, if you are tolerating the treatment well without significant side effects, you will come to the clinic once every 4 weeks. During these visits, you will have the following tests and procedures:

#### Day 1

- Physical examination
- Vital signs
- You will be given a supply of pazopanib each month with instructions on how to take the study drug and when to return to the doctor's clinic or office. Everyone who participates in this study will receive pazopanib in addition to the hormonal medication they are taking (either anastrozole or letrozole).
  - o For the rest of the study, you will take the study drug and either anastrozole or letrozole every day.
  - O You will take up to 4 tablets of pazopanib at least one hour before or two hours after a meal.
  - You should take both medications at about the same time each day.
  - o You will continue to obtain your hormonal treatment (anastrozole or letrozole) from your pharmacy as you have been prior to joining the study.

**Day 15, Day 28** 



- Physical examination
- Medical history
- Vital signs
- Blood tests (about 5-7 teaspoons) for the following
  - o For liver function tests you will have blood tests to monitor your liver function every 2 weeks during the first two months you are taking pazopanib
  - o To check for circulating tumor cells (if your blood test at screening showed that you have measurable circulating tumor cells) –Day 28 only, study test
- To measure your immune response –Day 28 only, study test
- ECG Day 28 only study test

If you are not experiencing any severe side effects, you will continue to be seen every 4 weeks until you stop taking pazopanib.

If you are experiencing severe side effects, you will continue to be seen every 2 weeks.

## Every 4 weeks and beyond

- Physical examination
- Vital signs
- Blood draw (about 3-5 teaspoons)
  - o For routine blood tests including liver function tests
  - o To check for circulating tumor cells (if you have measurable circulating tumor cells) at 12 weeks only study test
- Urine will be collected study test

## 12 weeks after starting pazopanib, and every 16 weeks thereafter

- ECG study test
- Disease assessment: CT or MRI or PET/CT or bone scan every 16 weeks unless your doctor requests that a scan be obtained sooner.

## When you are finished receiving pazopanib

You will return to the clinic within four weeks after you stop taking pazopanib. During this visit, you will have the following tests and procedures:

- Physical examination
- Vital signs
- Blood draw (about 3-5 teaspoons)
  - For routine blood tests
  - o To check for circulating tumor cells (if you have measurable circulating tumor cells) study test
- ECG study test
- Disease assessment CT, MRI, PET/CT or bone scan

IRB NUMBER: 11-07246 IRB APPROVAL DATE: 09/20/2017 IRB EXPIRATION DATE: 08/16/2018

**Study location:** All study procedures will be done at

UCSF – Mt. Zion

Helen Diller Family Comprehensive Cancer Center



## How long will I be in the study?

You will continue to receive pazopanib and your hormonal treatment as long as your disease does not progress or you do not have severe side effects, you experience any bad side effects, you decide to withdraw your consent to participate in this study, or the study is closed. If your cancer grows or if you begin another anti-cancer treatment, you will have to stop study treatment. After you are finished taking the treatment, the study doctor will ask you to visit the office for a follow-up exam within 4 weeks. The study team will contact you by phone each month for three months after your follow-up exam to see how you are doing.

## Can I stop being in the study?

Yes. You can decide to stop at any time. Tell the study doctor if you are thinking about stopping or decide to stop. He or she will tell you how to stop your participation safely.

It is important to tell the study doctor if you are thinking about stopping so any risks from stopping the pazopanib and hormonal treatment can be evaluated by your doctor. Another reason to tell your doctor that you are thinking about stopping is to discuss what follow-up care and testing could be most helpful for you.

The study doctor may stop you from taking part in this study at any time if he/she believes it is in your best interest, if you do not follow the study rules, or if the study is stopped.

## What side effects or risks can I expect from being in the study?

You may have side effects while on the study. Everyone taking part in the study will be watched carefully for any side effects. However, doctors don't know all the side effects that may happen. Side effects may be mild or very serious. Your health care team may give you medicines to help lessen side effects. If you develop side effects from the pazopanib, most should go away soon after you stop taking pazopanib. In some cases, side effects can be serious, long lasting, or may never go away.

You should talk to your study doctor about any side effects you experience while taking part in the study.



### Risks and side effects related to the study drug pazopanib

As of September 9, 2014, approximately 5875 patients and healthy volunteers had received pazopanib (either as monotherapy or in combination) out of more than 8600 patients enrolled in clinical studies of pazopanib. Pazopanib can cause side effects, although not everybody gets them. Some side effects can be life-threatening or fatal. The side effects below are those reported by patients who have taken pazopanib either in a clinical trial or as prescribed by their doctors. The side effects are listed according to the highest number of patients who had them in pazopanib studies, as very common, common, or uncommon. Not all side effects of pazopanib are known and further studies are under way. If you experience any side effects, please speak with your study doctor.

## Very common side effects occurring in more than 10% of patients include:

- diarrhea, feeling or being sick (nausea, vomiting, abdominal pain/discomfort)
- loss of strength and energy, weakness
- loss of appetite
- changes in hair color
- high blood pressure
- headache
- weight loss
- unusual hair loss or thinning
- a skin reaction or pain on the palms of the hands or soles of the feet (including tingling, numbness, pain, swelling or reddening)
- loss of skin pigment
- chest pain
- problems with taste
- mouth sores
- cough, shortness of breath
- dizziness
- skin rash
- muscle pain
- pain in the bones, muscles, ligaments, joints and tendons
- swelling caused by fluid in the hands, ankles, or feet
- slow heart rate

### Very common side effects that may show up in your blood tests:

increase in some substances (enzymes) produced by the liver. Patients over 60 years of age may be at greater risk of an increase of one of the enzymes, called ALT.

## Common side effects occurring in 1 - 10% of patients include:

- hoarse voice
- blurry vision
- indigestion



- nosebleeds
- blood in the urine
- low white blood cell counts neutropenia
- a decrease in the number of cells involved in blood clotting (thrombocytopenia)
- protein in the urine (a sign that kidneys are not working normally)
- under-active thyroid gland
- abnormal liver function
- increase in lipase (an enzyme from the pancreas)
- changes in heart's electrical conduction (QT-prolongation)
- temporary reduction in blood supply to the brain (mini-stroke)
- reduction of blood supply to the heart (angina)
- sudden collapse of the lung
- heart becomes less effective at pumping blood (cardiac dysfunction)
- chest pain, shortness of breath, leg pain, and swelling of the legs/feet. These could be signs of a blood clot in your body (thromboembolism). If the clot breaks off, it may travel to your lungs and this may be life threatening or even fatal
- severe bleeding in the lung
- heart attack
- chills
- rash, dry skin, nail disorder
- flatulence
- Inflammation of lining of the mouth
- Muscle spams

### Common side effects that may show up in your blood or urine tests:

- Increase in bilirubin (a substance produced by the liver)
- Increase in gamma-glutamyl transpeptidase (a liver enzyme)
- Decrease in albumin (a protein found in the blood)

## Uncommon side effects occurring in less than 1% of patients include:

- severe bleeding in digestive tract (stomach and intestine) and brain
- a dangerous rapid fluttering of the heart (Torsade de Points)
- hole in digestive tract which is called "perforation", which may require surgery to repair
- abnormal connection hole (perforation) in digestive tract
- stroke
- liver failure\*
- a sudden and severe rise in blood pressure (hypertensive crisis)
- inflammation of the pancreas
- Swelling of the brain that may be associated with high blood pressure, headache, loss of speech or vision, and/or seizure, which may be life threatening
- infections, with or without changes in white blood cells (cells that fight infection)

PAGE 8 OF 19

• separation or tear of the lining of the back part of the eye (retinal detachment or tear). This can result in blurry or impaired vision.

\*Two of the patients that received pazopanib died as a result of liver failure.

### Rare side effects (these may affect up to 1 in 1000 people):

• Blood clots accompanied by a decrease in red blood cells and cells involved in clotting. These clots may harm organs such as the brain and kidneys

### Other Risks of pazopanib

Neutropenia, thrombocytopenia, and palmar-plantar erythrodysaethesia syndrome were observed more frequently in patients of East Asian descent.

Studies in animals indicate that pazopanib may slow or stop bone growth. There is a possibility that pazopanib may affect bone growth in children, adolescents and young adults who are still growing.

During this study, blood tests will be checked to look for liver injury. People with liver injury may feel very tired or sick and not want to eat, have yellow skin or eyes, and they may also develop rash or fever. Let your doctor know if you have any of these symptoms, especially if your doctor says you have abnormal liver blood tests. If your doctor finds that your blood tests suggest liver injury that is not severe, your doctor may recommend you continue your study drug and may ask you to stop taking other drugs which may cause liver injury. Blood tests (about 1 teaspoon of blood per test) for possible liver injury will be repeated every week until you get better. If your blood tests get worse, your doctor may tell you to stop taking the study drug altogether. If you have a liver injury from the study drug, it will usually heal when the drug is stopped. It is possible that a small number of people may continue to have liver injury after they stop taking the study drug. There is a risk of liver failure, which could result in death.

If you are to have surgery, please speak with your doctor because pazopanib may affect wound healing.

#### Risks and side effects related to study procedures:

- **Safe Handling of Study Drug**: Handling pazopanib and having contact with any urine, feces or vomit from patients receiving pazopanib may pose some risk to you and your caregivers. To avoid exposure to pazopanib and any associated risks, you and your family members/caregivers will be educated by a member of the study team on how to safely handle, properly dispose of, and clean products that may be contaminated with pazopanib.
- **Blood drawing (venipuncture) risks:** Drawing blood may cause temporary discomfort from the needle stick, bruising, and infection.
- ECG risks: The adhesive on the leads may cause skin irritation including redness, itching, swelling or rash. These symptoms are generally mild and clear up on their own.

- Radiation (x-ray) risks: The amount of radiation you will be exposed to is relatively small. Such doses of radiation may be potentially harmful, but the risks are so small that they are difficult to measure. If you have already had many x-rays, you should discuss this with the researchers before agreeing to be in the study.
- CT scan risks: CT scans involve the risks of radiation (see above). In addition, if contrast material (iodine dye) is used, there is a slight risk of developing an allergic reaction, from mild (itching, rash) to severe (difficulty breathing, shock, or rarely, death). The contrast material may also cause kidney problems, especially if you are dehydrated or have poor kidney function. The study doctors will ask you about any allergies or related conditions before the procedure. If you have any of these problems, you may not be allowed to have a CT scan.

Having a CT scan may mean some added discomfort for you. In particular, you may be bothered by feelings of claustrophobia when placed inside the CT scanner, or by lying in one position for a long time. If contrast material is used, you may feel discomfort when it is injected into your vein. You may feel warm and flushed and get a metallic taste in your mouth. Rarely, the contrast material may cause nausea, vomiting or a headache

• MRI risks: Because the MRI machine acts like a large magnet, it could move iron-containing objects in the MRI room during your examination, which in the process could possibly harm you. Precautions have been taken to prevent such an event from happening; loose metal objects, like pocket knives or key chains, are not allowed in the MRI room. If you have a piece of metal in your body, such as a fragment in your eye, aneurysm clips, ear implants, spinal nerve stimulators, or a pacemaker, you will not be allowed into the MRI room and cannot have an MRI.

Having an MRI may mean some added discomfort for you. In particular, you may be bothered by feelings of claustrophobia and by the loud banging noise during the study. Temporary hearing loss has been reported from this loud noise. This is why you will be asked to wear ear plugs. At times during the test, you may be asked to not swallow for a while, which can be uncomfortable.

Because the risks to a fetus from MRI are unknown, pregnant women must not participate in this study.

Contrast agent (gadolinium) risks: A few side effects of gadolinium injection such as mild headache, nausea, and local pain may occur. Rarely (less than 1% of the time) low blood pressure and lightheadedness occurs. This can be treated immediately with intravenous fluids. Very rarely (less than one in one thousand), patients are allergic to gadolinium. These effects are most commonly hives and itchy eyes, but more severe reactions have been seen which result in shortness of breath.

Patients with severe kidney disease sometimes have a bad reaction to gadolinium contrast. The condition is called nephrogenic systemic fibrosis (NSF). It can cause skin to tighten or scar and can damage internal organs. Sometimes it can be life-threatening. There are no reports of

NSF in patients with normal kidney function. Before you have a MRI scan requiring an injection of gadolinium contrast, you will have a blood test in order to check the function of your kidneys. Based on your medical history and the results of the test, a doctor will decide whether it is safe for you to undergo the MRI scans.

- **PET/CT scan risks:** The PET scan exposes your body to radiation, see radiation risk above. The radiation levels come from a tracer which is a radioactive chemical injected into a vein in your arm. The tracer lets the doctor see how your cells are functioning and the radiation levels are very low. You may have an allergic reaction to the chemical used in the scan. For some patients, having to lie still on the scanning table for the length of the procedure may cause some discomfort or pain. After the scan your arm may be a little bit sore or have some redness where the IV was placed in your arm. The radioactive solution does not remain in your system for a long period of time. However, you should wait 2 hours before holding an infant or getting close to a pregnant woman to avoid exposing them to radiation. You should drink fluids after the scan to help remove the solution from your system.
- Bone scan risks: A bone scan is a diagnostic imaging test used to determine if your bone is damaged, either from cancer or from some other cause. The bone scan involves an injection, in the vein of your arm, of a radiotracer (radioactive compound that localizes in the bone). Most people do not experience any side effects from the radiotracer. The injection of the radiotracer may feel like a small sting, but there is no burning or other sensation as the radiotracer moves through your body. You will be exposed to a limited and medically acceptable dose of radiation during the procedure. There is always a slight risk of damage from being exposed to any radiation. If you are especially concerned with radiation exposure, please discuss this with your doctor.

Bone scan side effects are not common, and when encountered are usually mild, such as nausea and vomiting, or you may become uncomfortable lying still for the duration of the examination.

- **Tumor biopsy risks:** The general risks associated with this procedure are pain, discomfort, infection, bleeding and injury to organs nearby.
- Study drug combination risks: The side effects of the combination of pazopanib and anastrozole or letrozole are not yet known. It is possible that this combination of drugs will cause new or more serious side effects than taking these drugs separately. You will be monitored closely for side effects and your doctor may change your medications if it appears that this combination is causing serious side effects. You should tell your doctor about any side effects you experience while on this study. When additional information about side effects is known, you will be notified of any further study drug related effects.
- Study design risks: Since patients will be enrolled in a 2-step design, patients enrolled during the first step may receive a study drug that is not effective. Your study doctor will let you know which step you will be enrolled in.
- **Reproductive risks:** You should not become pregnant while on this study because the drugs in this study can affect an unborn baby. Women should not breastfeed a baby while on this

study. You will not be allowed to continue study treatment if you are or become pregnant. It is important to understand that you need to use birth control while on this study. Check with your study doctor about what kind of birth control methods to use and how long to use them. Some methods might not be approved for use in this study.

- Unknown Risks: The experimental treatments may have side effects that no one knows about yet. The researchers will let you know if they learn anything that might make you change your mind about participating in the study.
- For more information about risks and side effects, ask your study doctor.

## Are there benefits to taking part in the study?

Taking part in this study may or may not make your health better. While doctors hope the addition of pazopanib will be more useful against cancer compared to hormonal therapy alone, there is no proof of this. We do know that the information from this study will help doctors learn more about pazopanib as a treatment for breast cancer, and the benefit of combined pazopanib with hormonal treatment for breast cancer. This information could help future cancer patients. However, there is no guarantee that this will happen.

## What other choices do I have if I do not take part in this study?

Your other choices may include:

- Changing to a different hormonal therapy or starting chemotherapy.
- Getting treatment or care for your cancer without being in a study.
- Taking part in another study.
- Getting no treatment
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

If you decide not to participate in this study, your decision will not affect your medical care in any way.

Please talk to your doctor about your choices before deciding if you will take part in this study.

## Will my medical information be kept private?

We will do our best to make sure that the personal information in your medical record is kept private. However, we cannot guarantee total privacy. Your personal information may be given

out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- UCSF's Committee on Human Research
- Novartis Pharmaceuticals (the funder of the study) and their authorized agents
- UCSF Helen Diller Family Comprehensive Cancer Center (HDFCCC)
- The National Cancer Institute (NCI) and other government agencies, e.g., the Food and Drug Administration (FDA), involved in keeping research safe for people.
- The University of California
- Governmental agencies in other countries where the study drug may be considered for approval

Participation in research may involve a loss of privacy, but information about you will be handled as confidentially as possible. A medical record will be created because of your participation in this study. Your consent form and some of your research test results will be included in this record. Therefore, your other doctors may become aware of your participation. Hospital regulations require that all health care providers treat information in medical records confidentially.

## What are the costs of taking part in this study?

You and/or your health plan/insurance company will need to pay all of the costs of treating your cancer in this study, with the exception of tests done specifically for the study and not for treating your cancer. You and/or your insurance company will be responsible for paying for the costs of any procedures that are part of your standard medical care, such as your hormonal treatment, blood laboratory analyses, CT scans, MRI scans, PET scans, etc. Some health plans will not pay these costs for taking part in studies. Your study doctors or their clinical staff will obtain authorization from your insurance company prior to beginning your treatment. Taking part in this study may or may not cost you or your insurance company more than the cost of getting regular cancer treatment.

The study medication, pazopanib, will be provided to you at no charge. You will not be billed for any clinic visits or any of the tests required specifically by the study. These are procedures noted above as "study test" (such as blood draw for circulating tumor cells and to monitor your immune system, and collection of leftover tumor tissue) in this consent form.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's Web site at <a href="http://cancer.gov/clinicaltrials/understanding/insurance-coverage">http://cancer.gov/clinicaltrials/understanding/insurance-coverage</a>. You can print a copy of the "Clinical Trials and Insurance Coverage" information from this Web site.

Another way to get the information is to call **1-800-4-CANCER** (**1-800-422-6237**) and ask them to send you a free copy.



## Will I be paid for taking part in this study?

You will not be paid for taking part in this study.

## What happens if I am injured because I took part in this study?

It is important that you tell your study doctor, Hope Rugo, MD or her associates if you feel that you have been injured because of taking part in this study. You can tell the doctor in person or call him/her

**Treatment and Compensation for Injury:** If you are injured as a result of being in this study, the University of California will provide necessary medical treatment. The costs of the treatment may be billed to you or your insurer just like any other medical costs, or covered by the University of California depending on a number of factors. The University does not normally provide any other form of compensation for injury. For further information about this, you may call the office of the Committee on Human Research at 415-476-1814.

## What are my rights if I take part in this study?

Taking part in this study is your choice. You may choose either to take part or not to take part in the study. If you decide to take part in this study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your regular benefits. Leaving the study will not affect your medical care. You can still get your medical care from our institution

We will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

In the case of injury resulting from this study, you do not lose any of your legal rights to seek payment by signing this form.

## Who can answer my questions about the study?

You can talk to your study doctor about any questions, concerns, or complaints you have about this study. Contact your study doctor(s) (Hope Rugo, MD or her associates

If you wish to ask questions about the study or your rights as a research participant to someone other than the researchers or if you wish to voice any problems or concerns you may have about the study, please call the Office of the Committee on Human Research at 415-476-1814.



A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*

Please note: This section of the informed consent form is about an additional research study that is being done with people who are taking part in the main study. Participation in this extra research is voluntary, and if you choose not to donate your tissue for other analyses, it will in no way affect your care or participation in the main study.

You can say "yes" or "no" to the following study. Please mark and initial your choice.

## **About Using Tissue for Research**

We would like to ask that you have a tumor biopsy so we can use some of the tissue for additional research. If you agree, this tissue will be kept and may be used in research to learn more about cancer and other diseases. Please read the information sheet called "How Is Tissue Used for Research" to learn more about tissue research

The research that may be done with your tissue is not designed specifically to help you. It might help people who have cancer and other diseases in the future.

Reports about research done with your tissue will not be given to you or your doctor. These reports will not be put in your health record. The research will not have an effect on your care.

## Things to Think About

The choice to let us keep your biopsy tissue for additional research is up to you. No matter what you decide to do, it will not affect your care.

If you decide now that your tissue can be kept for research, you can change your mind at any time. Just contact us and let us know that you do not want us to use your tissue. Then any tissue that remains will no longer be used for research.

In the future, people who do research may need to know more about your health. While UCSF may give them reports about your health, it will not give them your name, address, phone number, or any other information that will let the researchers know who you are.

Sometimes tissue is used for genetic research (about diseases that are passed on in families). Even if your tissue is used for this kind of research, the results will not be put in your health records. If any commercial products are developed from the samples, you will not receive any reimbursement from any profits derived.

Your tissue will be used only for research and will not be sold. The research done with your tissue may help to develop new products in the future.

#### **Benefits**

The benefits of research using tissue include learning more about what causes cancer and other diseases, how to prevent them, and how to treat them. There may or may not be any direct benefit to you if you choose to participate in this optional research.

#### Risks

**Tumor biopsy risks**: The general risks associated with this procedure are pain, discomfort, infection, bleeding and injury to organs nearby.

The greatest risk to you is the release of information from your health records. We will do our best to make sure that your personal information will be kept private. The chance that this information will be given to someone else is very small.

## **Making Your Choice**

Please read each sentence below and think about your choice. After reading each sentence, put your initials in the "Yes" or "No" box. If you have any questions, please talk to your doctor or nurse, or call our research review board at IRB's phone number.

No matter what you decide to do, it will not affect your care.

1. My tissue may be kept for use in research to learn about, prevent, or treat cancer.

| YES | NO |
|-----|----|
|-----|----|

#### **CONSENT**

You have been given copies of this consent form and the Experimental Subject's Bill of Rights to keep.

You will be asked to sign a separate form authorizing access, use, creation, or disclosure of health information about you.

PARTICIPATION IN RESEARCH IS VOLUNTARY. You have the right to decline to participate or to withdraw at any point in this study without penalty or loss of benefits to which you are otherwise entitled.



| Date | Participant's Signature for Consent |
|------|-----------------------------------------------------------------|
| | Participant's Printed name |
| Date | Person Obtaining Consent |
| Date | Witness (only required if participant is a non-English speaker) |



## **Medications and Foods to Avoid**

## CC# 117513: Reversing Hormone Resistance in Advanced Breast Cancer with Pazopanib

The following is a list of medications to avoid while you are participating in this study. If you go to any medical visit, please take this list with you for the doctor's reference.

Before you begin treatment, Dr. Rugo or one of her associates will review all medications you are taking. Make sure you talk with Dr. Rugo before you start or stop taking any medications. This list contains only the most common drugs and food that are known to interact with the drugs used in this study. It is very important to discuss all medications that you are taking with your study doctor. This information will be reviewed at each study visit.

In addition to the listed medications, you should also avoid eating Seville (sour) oranges, grapefruit, starfruit and their juices.

## **Permitted Medications – Use with Caution**

| Generic Name | Brand Names ® | Generic Name | Brand Names ® |
|---|---|---|---|
| Amiodarone | Cordarone, Pacerone | Nevirapine | Viramune |
| Atomoxetine | Strattera | Oxcarbazepine | Trileptal |
| Bepridil | Vascor | Phenobarbital | Luminal |
| Carbamazepine | Carbatrol, Tegretol | Phenytoin | Dilantin |
| Clozapine | Clozaril, Fazaclo | Pimozide | Orap |
| Cortisone (>50mg) | | Pioglitazone | Actos |
| Cyclosporine | Sandimmune, Neoral,<br>Restatis, Gengraf | Prednisone (>10 mg) | Deltasone |
| Dexamethasone (>1.5 mg) | Decadron, Dexamethasone | Propafenone | Rythmol |
| Dihydroergotamine | DHE 45 | Quetiapine | Seroquel |
| Efavirenz | Sustiva | Quinidine | Cardioquin, Quinaglute |
| Ergonovine | | Rifabutin | Mycobutin |
| Ergotamine | Ergomar, Cafergot, Wigraine | Rifampin | Rifadin |
| Flecainide | Tambocor | Rifapentine | Priftin |
| Hydrocortisone (>40 mg) | Analpram HC, Carmol HC, Cortef, Cortenema | Risperidone | Risperdal |
| Lidocaine | Xylocaine | Sirolimus | Rapamune |
| Methylergonovine | Methergine | St John's Wort | |
| Methylprednisolone (>8 mg) | Medrol | Tacrolimus | Protopic, Prograf |
| Mexiletine | Mexitil | Warfarin | Coumadin, Jantoven |
| Modafinil | Provigil | | |

IRB NUMBER: 11-07246 IRB APPROVAL DATE: 09/20/2017 IRB EXPIRATION DATE: 08/16/2018

# **Prohibited Medications**

| Generic Name | Brand Names ® | Generic Name | Brand Names ® |
|----------------|----------------------|----------------|---------------|
| Amprenavir | Agenerase | Nefazodone | Serzone |
| Clarithromycin | Biaxin | Nelfinavir | Viracept |
| Fluconazole | Diflucan | Ritonavir | Norvir |
| Indinavir | Crixivan | Saquinavir | Invirase |
| Itraconazole | Sporanox | Telithromycin | Ketek |
| Ketoconazole | (oral forms only) | Troleandomycin | Tao |
| Lopinavir | (+ritonavir) Kaletra | Voriconazole | VFend |

Subjects should not receive other anti-cancer therapy [cytotoxic, biologic, radiation (other than leuprolide or other GnRH agonists)] while on treatment in this study.